CLINICAL TRIAL: NCT06828341
Title: A Single-arm, Open, Exploratory Clinical Study of Allogeneic CAR-T Cells in the Treatment of Relapsed/Refractory Brain Gliomas With Positive CD70 Expression
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: JIANG LONGWEI (Other)
Collaborators: Nanjing Kanghe Cell Gene Engineering Research Institute Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, JIANG LONGWEI, Associate Researcher, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SWZL20240122
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-05

CONDITIONS: Gliomas
Keywords: gliomas; car-t; allogeneic
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- allogeneic CAR-T targeting CD70 (Experimental): The enrolled patients will be received allogeneic CAR-T targeting CD70 that culutred from heathy adults. 1E6/kg CAR-T cells will be injected once from intrathecal.
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — allogeneic CAR-T targeting CD70 that cultured from heathy adults.

SUMMARY:
The goal of this clinical trial is to learn if allogeneic CAR-T cells can treat patients with advanced gliomas. The main questions it aims to answer are:

Evaluate the safety of allogeneic CAR-T cells in the treatment of advanced gliomas.

To evaluate the effectiveness of allogeneic CAR-T cells in the treatment of advanced gliomas and to study its immunological properties in patients.

DETAILED DESCRIPTION:
In this open, single-armed study, selected patients with advanced gliomas confirmed by Histopathology will be received allogeneic CAR-T cells treatment. First, their tumor specimen will be test to evaluate the expression of CD70.The patients with positive CD70 expression will be in enrolled.Then they will be received allogeneic CAR-T cells infusion cultured from heathy adults.

ELIGIBILITY:
Inclusion Criteria:

* 1) Agree to follow the study treatment plan and visit plan, voluntarily enroll, and sign the informed consent in writing; 2) Aged ≥18 years old on the day of signing the informed consent, regardless of gender; 3) Patients with recurrent/refractory glioma who have failed or cannot tolerate standard treatment and whose CD70 expression is confirmed by cytology or histology; 4) According to the results of immunohistochemistry test in a tertiary hospital (if historical tissue samples show CD70 positivity, no retest is required; if historical tissue samples show CD70 negative, a puncture biopsy is required) [historical archived tissue samples within 2 years are acceptable], the CD70 expression in the tumor site of the subject meets the positive standard, that is, ≥2+; 5) According to the RANO standard (Appendix 1), there is at least one evaluable or measurable lesion; 6) The expected survival period is ≥12 weeks; 7) The baseline Kanofsky performance score (Kanofsky performance score, KPS) score ≥ 70 points; 8) Subjects have adequate organ and bone marrow function and meet the following laboratory test standards: Bone marrow function: absolute neutrophil count (ANC) ≥ 1.5×109/L (1500/mm3); platelets (PLT) ≥ 90×109/L (1×105/mm3) (no blood transfusion or use of auxiliary white blood cells and platelets within 14 days before screening); White blood cell count ≥ 3.0×109/L (3000/mm3); Hemoglobin (HGB) ≥ 9.0 g/dL; Liver function: serum bilirubin (T-Bil) ≤ 1.5 times the upper limit of normal (ULN), Gilbert's syndrome (Gilbert's syndrome) (persistent or recurrent hyperbilirubinemia, manifested as elevated unconjugated bilirubin in the absence of evidence of hemolysis or liver pathology); patients without liver metastasis, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times ULN, patients with liver metastasis, ALT and AST ≤ 5 times ULN; Renal function: serum creatinine ≤ 1.5 times ULN, or creatinine clearance (Ccr) ≥ 50 mL/min (Ccr is calculated using the Cockcroft-Gault formula, see Appendix 5); Coagulation function: international normalized ratio (INR) ≤ 1.5 times ULN, activated partial thromboplastin time (APTT) ≤ 1.5 times ULN; 9) The investigator judges that the patient must have fully recovered from the previous treatment toxicity to ≤ Grade 1, except for the following situations: a. Alopecia; b. Pigmentation; c. Late toxicity caused by radiotherapy, which cannot be recovered by the investigator; d. Neurotoxicity of Grade 2 or below caused by platinum (CTCAE 5.0); Fertility-bearing male and female subjects of childbearing age must use effective contraceptive methods from the time they sign the informed consent until at least 6 months after CAR-T administration, and until 2 consecutive PCR tests show that there are no more CAR-T cells in the body. Women of childbearing age include premenopausal women and women within 2 years after menopause. Women of childbearing age must have a negative pregnancy test result within 7 days before the first dose.

Exclusion Criteria:

* 1) Patients who have received any treatment related to the CD70 target within 3 years; 2) Patients who have received any experimental drug treatment or used experimental devices within 28 days before CAR-T administration; 3) Patients who have received any systemic anti-tumor treatment within 28 days or 5 half-lives (whichever is longer) before CAR-T administration, including systemic chemotherapy, immunotherapy, hormone therapy (excluding glucocorticoids), targeted therapy, systemic immunomodulators (including but not limited to interferon, interleukin 2 and tumor necrosis factor), and received Chinese herbal medicine or Chinese patent medicine with anti-tumor effects within 14 days before CAR-T administration; 4) Patients who have received radiotherapy within three months before administration; 5) Patients who have received other non-CD70 target cell therapy products within two months before administration; 6) Patients who have received other cell therapy products in the past need to undergo RCL testing during the screening period, and patients with positive results in any test; 7) Patients who have received therapeutic doses of glucocorticoids within 14 days before CAR-T administration (however, physiological replacement doses of glucocorticoids are allowed, such as 10 mg/day prednisone or equivalent); 8) Patients who received oral or intravenous anticoagulation within 7 days before CAR-T cell administration; 9) Patients with other malignant tumors previously or concurrently, with the following exceptions: Carcinoma in situ that has been cured and has no signs of recurrence for at least 3 years before the study; The primary malignant tumor has been completely resected and in complete remission for ≥5 years. 10) History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 11) Those with immunodeficiency or autoimmune diseases, or those who need to use immunosuppressants; 12) Those who have received live vaccine immunization within 14 days before screening, or those who need to receive live vaccine immunization during the study; 13) Severe or uncontrollable systemic disease or any unstable systemic disease, including but not limited to uncontrolled hypertension, uncontrolled hyperglycemia, hepatic and renal dysfunction or metabolic diseases, central nervous system diseases, etc.; 14) Known severe cardiovascular disease, congenital long QT syndrome, torsades de pointes, myocardial infarction in the past 6 months, or arterial thrombosis, or unstable angina, or congestive heart failure of grade 3 or above (including grade 3) according to the New York Heart Association (NYHA) classification (see Appendix 3), or left ventricular ejection fraction (LVEF) <50%, QTc interval >450 ms for men and >470 ms for women ms; 15) Any one or both of the test results of Treponema pallidum antibody or human immunodeficiency virus (HIV) antibody are positive, cytomegalovirus (CMV) antibody IgM test is positive and CMV DNA titer is more than 2 times higher than the upper limit of normal value; Epstein-Barr virus antibody IgM test is positive and EBV DNA titer is more than 2 times higher than the upper limit of normal value; Hepatitis C virus antibody is positive and hepatitis C virus (HCV) RNA titer is more than 2 times higher than the upper limit of normal value, or active hepatitis B patients (defined as HBsAg positive and peripheral blood HBV DNA titer is more than 2 times higher than the upper limit of normal value); 16) Pregnant or lactating women; The researchers believe that the subjects have other conditions that may affect compliance or are not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of allogeneic T cells in the treatment of advanced giloma patients | 2 years
  The adverse events and severe adverse events will be evaluated.

SECONDARY OUTCOMES:
Evaluate the efficiency of allogeneic CAR-T cells in the treatment of advanced glioma patients. | 2 years
  The objective clinical response will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Shaochang, doctor, Study Chair — Jinling Hospital, China; GUO ZHIGANG, doctor, Study Director — Nanjing Normal University
Locations (1):
- Nanjing Jinling Hospital, China, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided